CLINICAL TRIAL: NCT03450044
Title: Immunogenicity and Safety of Autologous Dendritic Cells in Patients With Breast Cancer Treated With Neoadjuvant Chemotherapy.
Brief Title: Immunogenicity and Safety of DCs in Breast Cancer
Acronym: TEBICA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundación Salud de los Andes (Other)
Collaborators: Universidad Nacional de Colombia (Other); Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEBICA-001
Record Dates: First submitted 2018-02-12; First posted 2018-03-01 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer Female
Keywords: Chemotherapy; Breast Cancer; Dendritic cells; Immunotherapy; Doxorubicine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccinated (Experimental): Transfer of autologous dendritic cells interspersed with chemotherapy doses
  Interventions: Biological: Dendritic cells
- Control (No Intervention): Control patients who follow their basic treatment with chemotherapy with the A/C scheme

INTERVENTIONS:
Biological: Dendritic cells — Adoptive transfer of autologous DCs
  Arms: Vaccinated

SUMMARY:
This study aims to evaluate for the first time in Colombia the immunogenicity and safety of autologous DCs as enhancers of the immune response in patients with ductal breast cancer who, prior to surgical resection of the tumor, will receive neo-adjuvant chemotherapy with Doxorubicin and Cyclophosphamide. concomitantly with the transfer of autologous DCs. This clinical trial is based on the concept proposed in countries like France more than a decade ago, that chemotherapy or radiotherapy cause the tumor cells to release certain signals that favor the activation of the immune system against cancer. Therefore, the combined use of chemotherapy with vaccination with dendritic cells would provide the immune system with greater antitumor response capacity, taking advantage of the release of said signals to initiate a series of processes that would be reflected in the activation of T lymphocytes capable of destroying the remaining cells of the tumor. To determine the specificity of the response evoked by the adoptive transfer of autologous DCs, in each patient the degree of recognition of the tumor by the immune system before and after said procedure will be evaluated. These results will be compared with those of patients who participated in a control group.

Hypothesis Adoptive transfer of autologous DCs generated in vitro, in patients with stage IIA-IV breast cancer who receive neoadjuvant therapy with Doxorubicin and Cyclophosphamide, is a safe procedure that stimulates anti-tumor immune responses in treated patients.

Principal aim:

To evaluate the safety and immunogenicity of the use of DCs when used in patients with stage IIA-IV breast cancer in association with neo-adjuvant chemotherapy with Doxorubicin/Cyclophosphamide.

Specific aims:

* Generate immuno-competent dendritic cells in conditions of Good Clinical Practice and Good Laboratory Practices.
* Determine in each patient the immunological status of specific T lymphocytes against tumor antigens, before and after chemotherapy, in order to demonstrate whether the adoptive transfer of DCs favors the anti-tumor immune response.
* Register in patients with breast cancer in neo-adjuvant chemotherapy the class and frequency of adverse effects that could be generated as a result of the adoptive transfer of autologous DCs.

DETAILED DESCRIPTION:
The Fundación Salud de los Andes in the framework of a strategic alliance with the National University of Colombia has been working in the planning and development of a clinical trial in Colombia that promotes the search for new therapeutic alternatives for cancer patients. As a translational medicine project, it aims to make the laboratory findings available to the patient. This study explores the combination of immunotherapy (cell therapy) with chemotherapy, in order to obtain better results in the therapeutic management of tumors in patients with breast cancer.

Problem:

Breast cancer is a pathology that in recent years has increased vertiginously its incidence globally. Given the advanced state in which this tumor is usually diagnosed in our environment, the prognosis is seriously compromised, which has led to the current breast cancer represents a major public health problem in Colombia. The established therapies for the management of patients with this type of tumors such as chemotherapy, radio-therapy or surgery, are effective to reduce much of the established tumor mass, but fail to eliminate residual cancer cells, so - often - these treatments cannot prevent the recurrence of the disease. In addition to the above, the quality of life of the patients treated is strongly affected by the toxicity of these treatments on healthy tissues and their undesirable effects, which frequently affects poor adherence to treatment. That is why it is necessary to search for new therapeutic alternatives that are more specific to the tumor and that are better tolerated by patients. Due to the high specificity of the immune system for the recognition of tumors, different modalities of immune therapy for tumor control are currently being explored, which seek to enhance the performance of the patient's defense system so that a cytotoxic and memory response is established against them. tumor cells.

Type of study Clinical Trial Phase I / II.

Methodology:

Patients who attend the consultation due to their mammary pathology for the start of neo-adjuvant chemotherapy will be pre-selected to participate in the study. The participation of the volunteers will be subject to compliance with the inclusion and exclusion criteria defined for the study, as well as the signing of the informed consent. The participants will be randomly distributed into two groups.

PATIENT GROUPS As part of the clinical evaluation at the entrance of the study, a battery of laboratory tests (basic and specific to the trial) will be carried out. Subsequent to the corroboration of compliance with the inclusion criteria, patients will be randomly assigned to one of the two study groups: The first group (A) will be the negative control group, which includes patients who will receive only the standardized chemotherapy treatment for the pathology. The second group (B) will consist of those patients who were randomly selected to receive the adoptive transfer of mature autologous DCs in combination with the neo-adjuvant chemotherapy. In this way, the total of 30 patients will be distributed as follows: 15 patients for group A and 15 patients for group B.

The patients of group B will undergo an apheresis procedure in order to obtain a sample enriched in peripheral blood monocytes from which monocytes will be purified for the production of DCs. The generation of DCs will be carried out under strict conditions of Good Clinical Practices and Good Laboratory Practices.

The adoptive transfer will be carried out concomitantly with the neo-adjuvant chemotherapy treatment (eight and 15 days after chemotherapy dose for a total of 6 injections with autologous DCs).

In the period of application of the doses, a permanent clinical evaluation will be carried out to the patients, to register possible adverse effects (evaluation of the safety of the adoptive transfer of autologous DCs). The effect on the immune response of autologous DCs transferred to patients on chemotherapy vs. the effect on the immune response of chemotherapy without transfer, will be analyzed in each patient before and after chemotherapy using the state of the art of immunological techniques with which will measure the extent of anti-tumor CD8+ T cells expansion (evaluation of the immunogenicity of the adoptive transfer of autologous DCs).

Participating Institutions:

Fundación Salud de los Andes Research Group in Immunology and Clinical Oncology - GIIOC

National University of Colombia - Bogotá. School of Medicine Immunology and Translational Medicine Group Departments of Microbiology and Pathology

Other collaborating institutions:

Clínica del Seno Hospital Universitario Nacional Instituto Nacional de Cancerología Oncocare

ELIGIBILITY:
Inclusion criteria:

* Women between 30 and 65 years old.
* Patients who have histologically confirmed primary invasive ductal carcinoma of the breast.
* Patients who, at the time of their evaluation, present a breast cancer with TNM classification: IIA, IIB, IIIA, IIIB, IIIC or IV; in whom the breast-tumor relationship is not satisfactory for the surgical procedure, so that they will receive neo-adjuvant chemotherapy with Doxorubicin and Cyclophosphamide for at least 3 cycles.
* Patients who voluntarily agree to enter the proposed immunotherapy scheme.
* Absence of second malignant disease with the exception of a cervical carcinoma or a treated basal cell carcinoma.
* Normal blood, kidney function and hepatic function (neutrophil count 1000 / mm3, lymphocyte count 500 / mm3, hemoglobin 8mg / dl, and platelet count 150,000 / mm3, serum creatinine 1.5mg / dl, BUN 50mg / dl, aminotransferases 2 times of normal value and bilirubin 2.0mg / dl).
* Karnofsky higher than 70% or ECOG 0 to 1.
* Life expectancy greater than three months.
* Ability to understand informed consent.
* Have a weight greater than 50 Kilos at the time of apheresis.

Exclusion criteria:

* Patients who are pregnant or breast-feeding.
* Patients who have received some type of therapy as treatment for their tumor pathology in the breast, prior to the start of the trial (radiotherapy, chemotherapy, immunotherapy or gene therapy).
* Metastasis to the central nervous system at the time of inclusion in the study.
* Active autoimmune disease requiring treatment or history of autoimmune disease, which could be exacerbated by treatment. Patients with endocrine disease controlled by replacement therapy may be included, including thyroid disease, adrenal disease and vitiligo.
* Presence of a chronic or acute infection, such as HIV, viral hepatitis or tuberculosis, before or after the signing of the informed consent.
* Use of immunosuppressant within 4 weeks prior to the trial (eg corticosteroids), such as azathioprine, prednisone or cyclosporine A. The use of local steroids (topical, nasal or inhaled) may be acceptable.
* Patients with eczema, history of eczema or other eczematous skin disorders or those with acute or chronic exfoliative skin condition (eg atopic dermatitis, burns, impetigo, varicella zoster, severe acne or open wounds).
* Any disease that could interfere with the patient's ability to carry out the treatment (eg, Crohn's disease, ulcerative colitis or active diverticulitis, severe respiratory, cardiovascular, neurological, infectious disease or uncontrolled metabolic disease), including diseases of the psychiatric type.
* Clinically significant cardiomyopathy, which requires treatment.
* Splenectomized patients.
* Patients who do not receive the neo-adjuvant chemotherapy regimen with Doxorubicin and Cyclophosphamide for three cycles.
* Patients who have had an excisional biopsy.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Adverse effects | One year after innoculation
  Number of participants with treatment-related adverse events as associated with DCs inoculation assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Méndez, MD, Study Chair — CEO
Locations (1):
- Fundación Salud de los Andes, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banchereau J, Briere F, Caux C, Davoust J, Lebecque S, Liu YJ, Pulendran B, Palucka K. Immunobiology of dendritic cells. Annu Rev Immunol. 2000;18:767-811. doi: 10.1146/annurev.immunol.18.1.767. PMID 10837075
- [Background] Banchereau J, Palucka AK. Dendritic cells as therapeutic vaccines against cancer. Nat Rev Immunol. 2005 Apr;5(4):296-306. doi: 10.1038/nri1592. PMID 15803149
- [Background] Brossart P, Wirths S, Brugger W, Kanz L. Dendritic cells in cancer vaccines. Exp Hematol. 2001 Nov;29(11):1247-55. doi: 10.1016/s0301-472x(01)00730-5. PMID 11698120
- [Background] Butterfield LH, Ribas A, Dissette VB, Amarnani SN, Vu HT, Oseguera D, Wang HJ, Elashoff RM, McBride WH, Mukherji B, Cochran AJ, Glaspy JA, Economou JS. Determinant spreading associated with clinical response in dendritic cell-based immunotherapy for malignant melanoma. Clin Cancer Res. 2003 Mar;9(3):998-1008. PMID 12631598
- [Background] Chaput N, De Botton S, Obeid M, Apetoh L, Ghiringhelli F, Panaretakis T, Flament C, Zitvogel L, Kroemer G. Molecular determinants of immunogenic cell death: surface exposure of calreticulin makes the difference. J Mol Med (Berl). 2007 Oct;85(10):1069-76. doi: 10.1007/s00109-007-0214-1. Epub 2007 May 22. PMID 17891368
- [Background] Dauer M, Schad K, Herten J, Junkmann J, Bauer C, Kiefl R, Endres S, Eigler A. FastDC derived from human monocytes within 48 h effectively prime tumor antigen-specific cytotoxic T cells. J Immunol Methods. 2005 Jul;302(1-2):145-55. doi: 10.1016/j.jim.2005.05.010. PMID 15992809
- [Background] Dong Xda E, Ito N, Lotze MT, Demarco RA, Popovic P, Shand SH, Watkins S, Winikoff S, Brown CK, Bartlett DL, Zeh HJ 3rd. High mobility group box I (HMGB1) release from tumor cells after treatment: implications for development of targeted chemoimmunotherapy. J Immunother. 2007 Sep;30(6):596-606. doi: 10.1097/CJI.0b013e31804efc76. PMID 17667523
- [Background] Figdor CG, de Vries IJ, Lesterhuis WJ, Melief CJ. Dendritic cell immunotherapy: mapping the way. Nat Med. 2004 May;10(5):475-80. doi: 10.1038/nm1039. PMID 15122249
- [Background] Gabrilovich D. Mechanisms and functional significance of tumour-induced dendritic-cell defects. Nat Rev Immunol. 2004 Dec;4(12):941-52. doi: 10.1038/nri1498. PMID 15573129
- [Background] Kalinski P, Okada H. Polarized dendritic cells as cancer vaccines: directing effector-type T cells to tumors. Semin Immunol. 2010 Jun;22(3):173-82. doi: 10.1016/j.smim.2010.03.002. Epub 2010 Apr 20. PMID 20409732
- [Background] Mailliard RB, Wankowicz-Kalinska A, Cai Q, Wesa A, Hilkens CM, Kapsenberg ML, Kirkwood JM, Storkus WJ, Kalinski P. alpha-type-1 polarized dendritic cells: a novel immunization tool with optimized CTL-inducing activity. Cancer Res. 2004 Sep 1;64(17):5934-7. doi: 10.1158/0008-5472.CAN-04-1261. PMID 15342370
- [Background] Obeid M, Tesniere A, Ghiringhelli F, Fimia GM, Apetoh L, Perfettini JL, Castedo M, Mignot G, Panaretakis T, Casares N, Metivier D, Larochette N, van Endert P, Ciccosanti F, Piacentini M, Zitvogel L, Kroemer G. Calreticulin exposure dictates the immunogenicity of cancer cell death. Nat Med. 2007 Jan;13(1):54-61. doi: 10.1038/nm1523. Epub 2006 Dec 24. PMID 17187072
- [Background] Okada H, Kalinski P, Ueda R, Hoji A, Kohanbash G, Donegan TE, Mintz AH, Engh JA, Bartlett DL, Brown CK, Zeh H, Holtzman MP, Reinhart TA, Whiteside TL, Butterfield LH, Hamilton RL, Potter DM, Pollack IF, Salazar AM, Lieberman FS. Induction of CD8+ T-cell responses against novel glioma-associated antigen peptides and clinical activity by vaccinations with alpha-type 1 polarized dendritic cells and polyinosinic-polycytidylic acid stabilized by lysine and carboxymethylcellulose in patients with recurrent malignant glioma. J Clin Oncol. 2011 Jan 20;29(3):330-6. doi: 10.1200/JCO.2010.30.7744. Epub 2010 Dec 13. PMID 21149657
- [Background] Pinzon-Charry A, Maxwell T, Lopez JA. Dendritic cell dysfunction in cancer: a mechanism for immunosuppression. Immunol Cell Biol. 2005 Oct;83(5):451-61. doi: 10.1111/j.1440-1711.2005.01371.x. PMID 16174093
- [Background] Ramakrishnan R, Antonia S, Gabrilovich DI. Combined modality immunotherapy and chemotherapy: a new perspective. Cancer Immunol Immunother. 2008 Oct;57(10):1523-9. doi: 10.1007/s00262-008-0531-4. Epub 2008 May 17. PMID 18488219
- [Background] Romero P, Cerottini JC, Waanders GA. Novel methods to monitor antigen-specific cytotoxic T-cell responses in cancer immunotherapy. Mol Med Today. 1998 Jul;4(7):305-12. doi: 10.1016/s1357-4310(98)01280-5. PMID 9743992
- [Background] Zitvogel L, Apetoh L, Ghiringhelli F, Kroemer G. Immunological aspects of cancer chemotherapy. Nat Rev Immunol. 2008 Jan;8(1):59-73. doi: 10.1038/nri2216. PMID 18097448
- [Result] Bernal-Estevez D, Sanchez R, Tejada RE, Parra-Lopez C. Chemotherapy and radiation therapy elicits tumor specific T cell responses in a breast cancer patient. BMC Cancer. 2016 Aug 3;16:591. doi: 10.1186/s12885-016-2625-2. PMID 27484900
- [Result] Bernal-Estevez DA, Garcia O, Sanchez R, Parra-Lopez CA. Monitoring the responsiveness of T and antigen presenting cell compartments in breast cancer patients is useful to predict clinical tumor response to neoadjuvant chemotherapy. BMC Cancer. 2018 Jan 15;18(1):77. doi: 10.1186/s12885-017-3982-1. PMID 29334915
- [Derived] Bernal-Estevez DA, Ortiz Barbosa MA, Ortiz-Montero P, Cifuentes C, Sanchez R, Parra-Lopez CA. Autologous Dendritic Cells in Combination With Chemotherapy Restore Responsiveness of T Cells in Breast Cancer Patients: A Single-Arm Phase I/II Trial. Front Immunol. 2021 Aug 20;12:669965. doi: 10.3389/fimmu.2021.669965. eCollection 2021. PMID 34489928